CLINICAL TRIAL: NCT02727413
Title: Inflammatory and Vasoactive Mediator Profiles and Pathogen Characterization During Heart Valve Replacement Surgery
Brief Title: Inflammatory Mediator Profiles During Heart Valve Replacement Surgery
Acronym: Remove-Pilot
Status: Completed | Type: Observational
Sponsor: Jena University Hospital (Other)
Collaborators: Thermo Fisher Scientific, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: ZKS0071
Record Dates: First submitted 2016-03-23; First posted 2016-04-04 (Estimated); Last update posted 2019-06-24 (Actual); Status verified 2016-10

CONDITIONS: Infective Endocarditis; Valvular Heart Disease
MeSH Terms: conditions — Endocarditis; Heart Valve Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Infective endocarditis: Blood sample collection and assessment of signs of organ dysfunction in patients diagnosed with infective endocarditis in accordance with Duke criteria and scheduled for valve surgery
  Interventions: Procedure: Blood sample collection; Other: Assessment of signs of organ dysfunction
- Valvular heart disease: Blood sample collection and assessment of signs of organ dysfunction in patients diagnosed with valvular heart disease, with no signs of infection, scheduled for valve replacement surgery
  Interventions: Procedure: Blood sample collection; Other: Assessment of signs of organ dysfunction

INTERVENTIONS:
Procedure: Blood sample collection — Drawing of 10 ml blood at inclusion, at the time of CPB connection, 60 min under CPB, at the time of CPB disconnection, 6, 24 and 48 hours post-surgery
Other: Assessment of signs of organ dysfunction — Assessment of signs of organ dysfunction based on medical data prior to surgery, 24 and 48 hours post-surgery, and at the time of ICU discharge
  Other Names: SOFA score

SUMMARY:
The study aims at the comparative examination of pre-, intra- and post-operative release profiles of inflammatory and vasoactive mediators in patients undergoing heart valve surgery under cardiopulmonary bypass (CPB) due to either infectious endocarditis or degenerative valvular heart disease. Specific attention will focus on the distinction between mediator release associated with infection and that resulting from CPB. Concomitantly identification and characterization of infectious pathogens in the circulation and in valvular samples will be carried out, together with the search for resistance-coding transcripts.

DETAILED DESCRIPTION:
Exaggerated release of inflammatory mediators and endogenous vasoactive substances resulting from the coincident infection and surgical stress plays a role in post-operative organ failure and altered immune defense, thus contributing to unfavorable post-operative outcome.

Cardiopulmonary bypass (CPB) itself, even in the absence of IE, has been shown to modify cytokine and vasoactive mediator release and may cause organ failure. Tracing of release profiles of inflammatory cytokines and vasoactive mediators and their correlation with postoperative organ dysfunction in cardiac surgery for IE or non-IE patients aims at the assessment of the prognostic validity of these biomarkers and the evaluation of measures for their pro-active clearance during the surgical intervention.

Induction of inflammatory mediators and their temporal release profile may vary depending on the involved pathogens, which cannot be always identified by conventional techniques (blood culture). Since it is conceivable that identification of the involved pathogen could explain differences in cytokine secretory patterns in IE, use of advanced molecular technologies (NGS) will support the clarification of such relations. Analysis of transcripts encoding inflammatory and vasoactive mediators in blood cells will enable the surveillance of temporal oscillations in their profiles during the observation time frame. Transcriptome analysis of identified putative pathogens can also disclose features of antibiotic resistance.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent
* age > 18
* confirmed diagnosis of infective endocarditis or valvular heart disease
* scheduled surgical Intervention with CPB use

Exclusion Criteria:

* glucocorticoid dosage above Cushing threshold
* severe neutropenia (below 1000/mm3)
* immunosuppression or immunomodulatory therapy
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with infective endocarditis or valvular heart disease, undergoing cardiac surgery with cardiopulmonary bypass
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of Procalcitonin | 24 h before surgery - connection/disconnection of CPB - 24 and 48 h post-surgery
  Plasma levels of Procalcitonin over time
Area under the plasma concentration versus time curve (AUC) of C-reactive Protein (CRP) | 24 h before surgery - connection/disconnection of CPB - 24 and 48 h post-surgery
  Plasma Levels of CRP over time
Area under the plasma concentration versus time curve (AUC) of Endothelin 1 | 24 h before surgery - connection/disconnection of CPB - 24 and 48 h post-surgery
  Plasma Levels of Endothelin 1 over time
Area under the plasma concentration versus time curve (AUC) of Tumor Necrosis Factor (TNF) alpha | 24 h before surgery - connection/disconnection of CPB - 24 and 48 h post-surgery
  Plasma Levels of TNF alpha over time
Area under the plasma concentration versus time curve (AUC) of Interleukin (IL) 1beta | 24 h before surgery - connection/disconnection of CPB - 24 and 48 h post-surgery
  Plasma Levels of IL 1beta over time
Area under the plasma concentration versus time curve (AUC) of Interleukin (IL) 6 | 24 h before surgery - connection/disconnection of CPB - 24 and 48 h post-surgery
  Plasma Levels of IL 6 over time
Area under the plasma concentration versus time curve (AUC) of Interleukin (IL) 10 | 24 h before surgery - connection/disconnection of CPB - 24 and 48 h post-surgery
  Plasma Levels of IL 10 over time
Area under the plasma concentration versus time curve (AUC) of Interleukin (IL) 18 | 24 h before surgery - connection/disconnection of CPB - 24 and 48 h post-surgery
  Plasma Levels of IL 18 over time

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of pro-Adrenomedullin | 24 h before surgery - connection/disconnection of CPB - 24 and 48 h post-surgery
  Plasma Levels of pro-Adrenomedullin
Area under the plasma concentration versus time curve (AUC) of pro-Arginine vasopressin | 24 h before surgery - connection/disconnection of CPB - 24 and 48 h post-surgery
  Plasma Levels of pro-Arginine vasopressin
Area under the plasma concentration versus time curve (AUC) of pro-Atrial natriuretic peptide | 24 h before surgery - connection/disconnection of CPB - 24 and 48 h post-surgery
  Plasma Levels of pro-Atrial natriuretic peptide
SOFA Score | 24 h before and 24 and 48 h after surgical intervention
  Changes in SOFA scores after surgery, as compared to pre-surgery baseline
Renal replacement therapy | Over 7 days following surgery
  Use and duration of renal replacement therapy
Concomitant medication | During and 48 h upon completion of surgical intervention
  Cumulative doses of applied vasopressors, corticosteroids and prostaglandins
In-hospital mortality | 30 days after surgery
  Post-surgical mortality over 30 days

OTHER OUTCOMES:
Pathogen genotyping | Before and during intervention at the heart valve
  Identification of circulating pathogens
Resistance transcripts | During intervention at the heart valve
  Abundance of bacterial transcripts encoding antibiotic resistance in blood

CONTACTS AND LOCATIONS:
Overall Officials: Frank M Brunkhorst, MD, Study Chair — Jena University Hospital
Locations (1):
- Center for Clinical Studies, Jena University Hospital, Jena, Thuringia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Diab M, Tasar R, Sponholz C, Lehmann T, Pletz MW, Bauer M, Brunkhorst FM, Doenst T. Changes in inflammatory and vasoactive mediator profiles during valvular surgery with or without infective endocarditis: A case control pilot study. PLoS One. 2020 Feb 3;15(2):e0228286. doi: 10.1371/journal.pone.0228286. eCollection 2020. PMID 32015566